CLINICAL TRIAL: NCT03226717
Title: Effects of Direct Antiviral Agents on Hepatitis C Virus Arthropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin abd elazim mohamed turkey, principle investigator., Assiut University
Other Study IDs: HCVDAV
Record Dates: First submitted 2017-06-18; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Antiviral Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hepatitis C patients: Antiviral agents (sofosbuvir,daclatasvir,ribavirin) will be given to hepatitis C patients with arthropathy.
  Interventions: Drug: Antiviral agents

INTERVENTIONS:
Drug: Antiviral agents — combination therapy consists of Sofosbuvir,daclatasvir and ribavirin

SUMMARY:
The prevalence of HCV infection in Egypt is 14.7%. HCV is both a hepatotropic and a lymphotropic virus, it may exert a chronic stimulus on the immune system with both T and B lymphocyte alterations. In addition to cryoglobulinaemic vasculitis, HCV may trigger different immune-mediated extrahepatic disorders. A variable combination of HCV with other unknown enviromental and/or hostgenetic cofactors may lead to different clinical phenotypes that characterise HCV syndrome. Patients who have HCV -related arthropathy are accounted for by 2 clinical subsits: Rheumatoid-like arthritis and Cryoglobulin-related arthritis. Patients with mild arthritis, conservative manegement using analgesics with anti- inflammatory activity is recommended. In patients who have contraindications to their use, short term low dose prednisone is an option. In HCV infection with concomitant RA, ACR guidelines published in 2008 provided recommendations pertaining to these of DMARDs that are based on the severity of liver disease using the child- pugh- turcotte classification. For patients with severe cryoglobulinaemia such as severe debilitating disease or systemic in improvement, a combination of immunosuppressive and antiviral therapy is preferred. It has been found that antiviral therapy with interferon immunosuppressive and antiviral therapy is preferred. It has been found that antiviral therapy with interferon improves the musculoskeletal manifestations in HCV arthropathy. The DIrect antiviral agents seems very promising in treatment of HCV arthropathy. As HCV genotype 4 is the most common genotype in Egypt, the effective optional antiviral agents are sofosbuvir, daclatasvir, ledipasvir, paritaprevir, velpatasvir, ombitasvir and simeprevir.

ELIGIBILITY:
Inclusion Criteria:

* Antiviral patients with arthropathy concomitant HCV (proved by PCR testing).

Exclusion Criteria:

* patients with child-pugh B and child-pugh C decompensated cirrhosis.
* patients more that 60 years.
* patients with chronic infection e.g.(pulmonary T.B).
* patients with organ failure e.g.( heart failure, respiratory failure).
* patients with CKD with GFR lead that 60 ml/ ministry/1.73m2.
* patients on immunosuppressive agents.
* patients with HBV- coinfection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with hepatitis C virus
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-10 (Estimated); Primary Completion 2017-09-10 (Estimated); Study Completion 2017-12-10 (Estimated)

PRIMARY OUTCOMES:
rate of Improvement of manifestations of arthropathy | 3_6 months
  Improvement of manifestations of arthropathy in hepatitis C patients after treatment by assessment through pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- yasmin AbdElazim Mohamed Turkey, Asyut, Egypt